CLINICAL TRIAL: NCT00718185
Title: The Pharmacokinetics and Pharmacodynamics of Sildenafil in Pediatric and Adult Patients
Brief Title: Pharmacokinetics and Pharmacdynamics of Sildenafil
Status: Terminated | Type: Observational
Why Stopped: Similar study completed.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-11-5636
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2010-02

CONDITIONS: Pulmonary Hypertension
Keywords: Sildenafil; Pediatrics
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients receiving sildenafil as standard of care
  Interventions: Procedure: Obtain blood specimens

INTERVENTIONS:
Procedure: Obtain blood specimens — Obtain blood samples at multiple timepoints.

SUMMARY:
The study is being done to investigate what happens to sildenafil in the body and how long it takes to get rid of this drug. Understanding how long the drug stays in the body and how it is changed by the body will help doctors determine the best dose. We also want to learn how well the medicine works based on the size of the dose or amount in the bloodstream.

DETAILED DESCRIPTION:
There is no data regarding sildenafil drug disposition in infants and children with pulmonary hypertension. Sildenafil is used at The Children's Hospital of Philadelphia for the treatment of pulmonary hypertension. Patients receiving sildenafil as standard of care will be approached for consent.

ELIGIBILITY:
Inclusion Criteria:

* Receive enteral sildenafil as standard of care
* > 28 days to >18 years of age
* Informed consent/assent

Exclusion Criteria:

* Parents/guardians and/or subjects who, in the opinion of the investigator, may be noncompliant with study schedules or procedures.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants, Children, and Adults receiving sildenafil as standard of care for the treatment of pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To define the PK of sildenafil administered as standard of care in infants with pulmonary hypertension | predose, .5mins after dose, 2-4 hrs after dose, and 5-7 hrs after dose

SECONDARY OUTCOMES:
To describe the PD effects of sildenafil administered as standard of care in infants and children with pulmonary hypertension. | Multiple time points throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States